CLINICAL TRIAL: NCT07096934
Title: A Prospective, Randomized, Controlled Trial to Evaluate the Safety and Efficacy of CYWC628 (Human Dermal Fibroblast Spheroids) for the Treatment of Refractory Diabetic Foot Ulcers Compared With Standard of Care
Brief Title: Controlled Trial to Evaluate the Safety and Efficacy of CYWC628 (Human Dermal Fibroblast Spheroids) for the Treatment of Refractory Diabetic Foot Ulcers Compared With Standard of Care
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FibroBiologics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYWC628-CLIN-001
Record Dates: First submitted 2025-07-09; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: DFU; Diabetic ulcers; diabetic wounds; diabetic foot ulcers; chronic wounds; chronic ulcers; non-healing wounds
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Approximately 120 participants will be randomized in parallel to one of the following treatment groups (40 participants per group):
  1. SoC + Low dose CYWC628
  2. SoC + High dose CYWC628
  3. SoC only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of Care (Active Comparator): Standard of care used for the treatment of diabetic foot ulcers once weekly for up to 12 weeks.
  Interventions: Other: Standard of Care (SOC)
- SoC + Low dose CYWC628 (Experimental): standard of care (SoC) + low dose CYWC628 applied once weekly to diabetic foot ulcer (DFU) for up to 12 weeks:
  Interventions: Biological: SoC + Low dose CYWC628
- SoC + High dose CYWC628 (Experimental): standard of care + high dose CYWC628 applied once weekly to diabetic foot ulcer (DFU) for up to 12 weeks:
  Interventions: Biological: SoC + High dose CYWC628

INTERVENTIONS:
Other: Standard of Care (SOC) — The participant's DFU will be sharply debrided (as needed), dressed with SoC and offloaded.
  Arms: Standard of Care
Biological: SoC + Low dose CYWC628 — The participant's DFU will be sharply debrided (as needed), dressed with SoC and offloaded. Low dose CYWC628 applied once weekly to diabetic foot ulcer (DFU) for up to 12 weeks
  Arms: SoC + Low dose CYWC628
Biological: SoC + High dose CYWC628 — The participant's DFU will be sharply debrided (as needed), dressed with SoC and offloaded. High dose CYWC628 applied once weekly to diabetic foot ulcer (DFU) for up to 12 weeks
  Arms: SoC + High dose CYWC628

SUMMARY:
This is a prospective, multicentre, randomized clinical trial evaluating the safety, tolerability, and efficacy of up to 12 weeks treatment with SoC + low- or high-dose CYWC628 in treating DFU, compared to SoC only.

DETAILED DESCRIPTION:
This is a prospective, multicentre, randomized clinical trial evaluating the safety, tolerability, and efficacy of up to 12 weeks treatment with SoC + low- or high-dose CYWC628 in treating DFU, compared to SoC only.

Period 1:

After providing voluntary, written informed consent, participants will undergo screening assessments according to the schedule of assessments (SOA). The participant's DFU will be sharply debrided (as needed), dressed with SoC and offloaded. If there is evidence of infection, a skin pathogen test will be performed and topical or systemic antibiotic or antifungal may be administered until the infection is cleared or is at a level defined as acceptable in the eligibility criteria.

After the Screening visit (or the visit at which any DFU infection is deemed cleared or is at a level defined as acceptable in the eligibility criteria), the participant will return two (2) weeks later to confirm eligibility. If the DFU wound area has not decreased in size ≥30% and the participant remains eligible, they will be randomized on Day 1 to one of 3 treatment groups: SoC + low dose CYWC628, SoC + high dose CYWC628, or SoC only.

The treatment period is comprised of weekly visits for allocated study treatment for up to 12 weeks (i.e., up to 12 treatments). At each visit, the DFU will be assessed by the Investigator and measured using the eKare inSight® electronic image capture application, and ABI determined. Vital signs and clinical laboratory testing will be performed at each study visit, from Day 1 until the Week 12 visit or the visit at which the DFU is deemed healed by the Investigator (whichever visit occurs first). Adverse events and concomitant medications/therapies will be recorded at each visit.

The Safety Review Committee (SRC) will review the safety data from the first 2 weeks treatment of the first 20 randomized participants (sentinel group), i.e., data from Day 1, Week 1 and Week 2 visits. If safety and tolerability is confirmed as acceptable, enrolment of the remaining participants will proceed. An interim analysis will be performed when at least 28 randomized participants per treatment group have completed the Week 6 visit, to assess primary safety and efficacy endpoints at Week 6.

Period 1 participants whose DFU heals within the 12-week treatment period (regardless of treatment) will attend 2 follow-up visits 2 weeks apart to confirm healing and attend the end of study visit (EOS) at 6 months post-last treatment. At each follow-up visit, any recurrence of the DFU at the same site will be assessed and recorded.

Period 1 participants randomized to SoC + CYWC628 whose DFU does not heal within 12 weeks, and participants randomized to SoC only whose DFU does not heal within 12 weeks and do not continue with Period 2 treatment with SoC + CYWC628, will revert to their treating physician's care for DFU. Safety follow-up visits for SoC + CYWC628-treated participants with non-healed DFU will be performed at Weeks 14 and 16, with the Week 16 visit considered the EOS for these participants. Safety follow-up visits for SoC only-treated participants with non-healed DFU will be performed at the Week 16 visit only, with this visit considered the EOS for these participants.

Period 2:

Period 1 participants randomized to SoC only whose DFU does not heal within the Period 1 12-week treatment period will be offered up to 12 weeks treatment with SoC + CYWC628 if remaining eligible and at the discretion of the Investigator.

Before participants receive Period 2 treatment with SoC + CYWC628, eligibility must be re-confirmed (Period 1 Week 12 visit assessments may be used with addition of toe systolic pressure measurement; serology and ECG not required unless considered necessary by Investigator). The same 2-week period required between Period 1 Screening and Day 1 randomization will also apply between the Period 1 Week 12 visit and first administration of Period 2 SoC + CYWC628 treatment. Procedures for treatment for infected DFU described for Period 1 Screening will also be applied in Period 2. Eligible participants will receive a dose of CYWC628 if a safe and effective dose has been determined from the interim analysis. Treatment with SoC + CYWC628 and follow-up visits in Period 2 will be as described for Period 1, except that the EOS will be performed 4 weeks after DFU deemed healed by the Investigator (or Period 2 Week 16 visit if unhealed in 12 weeks). Period 2 will not proceed if not approved by the SRC.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 80 years inclusive at time of informed consent.
2. Diagnosed/confirmed Type 1 or 2 diabetes mellitus.
3. Presence of diabetic foot ulcer (DFU) at or below the level of the malleolus that is confined to one anatomical site and without exposure of bone and/or joint capsule.
4. DFU Wagner Grade 1 or 2.
5. DFU present for 12 to 52 weeks at time of Screening.
6. DFU cross-sectional area of 50 to 1000 mm2 at Screening and Day 1.
7. Resting ankle brachial index (ABI) ≥0.6 and ≤1.2, or toe pressure >30 mmHg.
8. HbA1c <9%.
9. Non-infected DFU (i.e., Infectious Diseases Society of America [IDSA] International Working Group on the Diabetic Foot [IWGDF] Classification 1/Uninfected) OR, at the discretion of the Investigator, DFU infection of IWGDF/IDSA Classification 2/Mild, at least within 2 weeks before and on Day 1.

   At the discretion of the Investigator, if the DFU infection is IWGDF/IDSA Classification 3/ Moderate at Screening, the Screening period may be extended to allow time to reduce the infection to IWGDF/IDSA Classification 2/ Mild or 1/ no infection at least 2 weeks before randomization on Day 1. Otherwise, DFU infection of IWGDF/IDSA Classification ≥3 and/or any infection involving bone (osteomyelitis), is exclusionary.

   If there is evidence of infection during the Screening period (i.e., only IWGDF/IDSA Classification 2/ Moderate or 3/ Severe), the following will be performed:
   * A skin pathogen test;
   * Treatment with systemic or topical antibiotic or antifungal as deemed required by the Investigator. Systemic treatment must have ceased at least 5 days before Day 1. Ongoing topical antibiotic or antifungal treatment after randomization is permitted;
   * Continue treatment of IWGDF/IDSA Classification 3/ Moderate infection as required until reduced to IWGDF/IDSA Classification 2/ Mild or 1/ no infection by at least 2 weeks before Day 1
   * Sharp debridement of any further necrotic tissue, slough, or biofilm as needed.
10. If participant of child bearing potential, must have a negative serum pregnancy test at screening and negative urine pregnancy test pre-first treatment on Day 1, and must agree to remain sexually abstinent, or use medically effective contraception (refer to Appendix 11.1), or have a partner who is sterile or same-sex, from Screening until at least 60 days after the last dose of study treatment. Males must not be planning to father children or donate sperm for the duration of the study and for at least 90 days after the last dose of study product.
11. Understands and is able and willing to participate and comply with study requirements including attending study visits and follow-up.

Exclusion Criteria:

1. The DFU had been previously treated, or is being treated, with growth factors, stem cells, or any equivalent preparation within 8 weeks before Screening.
2. Enrolment in another interventional clinical foot ulcer healing trial within 4 weeks before Screening, or participation in any other interventional research study within 8 weeks before screening.
3. Additional wound(s) within 3 cm of the study target wound.
4. History of conditions that may impair wound healing in the opinion of the Investigator, for example, autoimmune disorders, renal failure patients on dialysis, or medications that impair the healing process. .
5. DFU with exposure of bone and/or joint capsule.
6. Active osteomyelitis, cellulitis, soft tissue infection, or Charcot's arthropathy present on the affected foot or limb containing the DFU, or DFU infection IWGDF/IDSA Classification 4/ Severe, or DFU infection IWGDF/IDSA Classification 3/ Moderate at Screening that cannot be reduced to Classification 2/ Mild or Classification 1/ No infection with treatment.
7. Active healing and reduction of wound area ≥30% during the two-week period before Day 1.
8. Known allergy to topical dressings, any of the study treatment components, and/or to gentamicin or other aminoglycosides.
9. Use of systemic antibiotics or antifungals for treatment of or prophylaxis for DFU infection within 5 days before Day 1, and/or if such use is considered by the Investigator likely to be required during the study treatment period. Systemic antibiotic or antifungal use for other indications is not exclusionary.
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer considered treated and cured) within 5 years of screening, regardless of whether there is no evidence of local recurrence or metastasis. Basal cell carcinomas of the skin are also exclusionary if diagnosed within 6 months before screening. If there is suspicion of skin cancer, a biopsy may be performed during screening for confirmation.
11. Pregnant or breastfeeding, or a male participant planning to father children or donate sperm during the study and for 90 days after last dose of study treatment.
12. Current smoker of tobacco products and/or active user of nicotine replacement products including but not limited to nicotine gum, patches, or vaping.
13. Current alcohol misuse as determined by the Investigator, and/or positive alcohol breath test at screening or pre-first treatment (no re-test permitted).
14. Substance use disorder of any severity as determined by the Investigator, including any use of illicit drugs or other addiction which might interfere with the ability to comply with study procedures in the opinion of the Investigator; positive urine drug test at screening or pre-first treatment (tricyclic antidepressants, opioids, cannabidiols [CBDs] and benzodiazepines are not exclusionary if prescribed by a physician and consistent with medical history). One re-test permitted for urine drug test where justified in the opinion of the Investigator (e.g., false positive suspected).
15. Any other condition or situation that, in the opinion of the Investigator, would compromise the participant's ability to comply with study requirements.
16. Known history of poor compliance with medical treatments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate Adverse events, including severity grading using Common Terminology Criteria for Adverse Events (CTCAE v5.0), and relationship to treatment | from enrollment to the end of the treatment at 12 weeks
  Evaluate the safety and tolerability of Standard of Care (SoC) + CYWC628 in patients with diabetic foot ulcer (DFU) as compared to SoC only.
  • Adverse events, including severity grading using Common Terminology Criteria for Adverse Events (CTCAE v5.0), and relationship to treatment.
Evaluate proportion of participants with complete wound closure by 12 weeks after commencing study treatment or SoC | from enrollment to the end of the treatment at 12 weeks
  Evaluate the efficacy of SoC + low dose and high dose CYWC628 in wound healing of DFU, compared with SoC only.
  Proportion of participants with complete wound closure by 12 weeks after commencing study treatment or SoC. Complete wound closure is defined as 100% re-epithelialization with no wound drainage, as determined by the Investigator, observed at 2 visits 2 weeks apart
Evaluate percentage area reduction (PAR) of the DFU wound during the 12 week treatment period. | from enrollment to the end of the treatment at 12 weeks
  Evaluate the safety and tolerability of Standard of Care (SoC) + CYWC628 in patients with diabetic foot ulcer (DFU) as compared to SoC only.
  Percentage area reduction (PAR) of the DFU wound during the 12 week treatment period.

SECONDARY OUTCOMES:
Evaluate the treatment time to complete wound healing of DFU by SoC + CYWC628, compared to SoC only | from enrollment to the end of the treatment at 12 weeks
  To assess the treatment time of wound healing of DFU by SoC + CYWC628, compared to SoC only.
  Time (days) to complete wound closure after commencing SoC + CYWC628 treatment or SoC only
Complete wound closure and PAR in SoC patients offered treatment at the end of the 12 week primary outcome | from enrollment to the end of the treatment at 12 weeks
  participants randomized to SoC only whose DFU does not heal within the Period 1 12-week treatment period will be offered up to 12 weeks treatment with SoC + CYWC628 if remaining eligible and at the discretion of the Investigator. Proportion of participants with complete wound closure by 12 weeks after commencing SoC + CYWC628.
  Percentage area reduction (PAR) of the DFU wound during the 12 week treatment period with SoC + CYWC628.
Evaluate DFU recurrence rate in patients with successful wound healing within 12 weeks of study treatment | DFU at the same site within 6 months of original complete wound healing (last treatment). Time to recurrence of DFU within 6 months of complete wound healing (last treatment).
  To assess the recurrence rate of treated DFU at the same site, after successful wound healing within 12 weeks of study treatment (Period 1 only).
  Proportion of participants reporting a recurrence of DFU at the same site within 6 months of original complete wound healing (last treatment).
  Time to recurrence of DFU within 6 months of complete wound healing (last treatment).
Evaluate improvement in vascularization in patients administered SoC + CYWC628 | from enrollment to the end of the treatment at 12 weeks
  To assess if DFU treatment with SoC + CYWC628 improves vascularization and thereby circulation.
  Ankle brachial index (ABI) measurements compared to baseline. At each treatment visit, proportion of participants with ABI in each of categories: normal (1.0-1.4), borderline (0.91-0.99), abnormal (PAD) (<0.90), Non-compressible arteries (>1.40).

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Khoja Chief Scientific Officer, Ph.D., Principal Investigator — FibroBiologics

IPD SHARING:
Plan to Share IPD: Yes
we will share de-identified data collected for the primary and secondary outcomes of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the end of the study and after the publication of the data.